CLINICAL TRIAL: NCT02223026
Title: Relative Bioavailability of a 2.5 mg Linagliptin / 1000 mg Metformin Fixed Dose Combination Tablet Administered With and Without Food to Healthy Male and Female Subjects in an Open, Randomised, Single-dose, Two-way Crossover, Phase I Trial
Brief Title: Relative Bioavailability of a Linagliptin+Metformin Fixed Dose Combination Tablet Administered With and Without Food to Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.4
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (2):
- Linagliptin/metformin fed (Experimental)
  Interventions: Drug: Linagliptin/metformin FDC; Other: high-fat, high caloric meal
- Linagliptin/metformin fasted (Active Comparator)
  Interventions: Drug: Linagliptin/metformin FDC

INTERVENTIONS:
Drug: Linagliptin/metformin FDC
Other: high-fat, high caloric meal
  Arms: Linagliptin/metformin fed

SUMMARY:
Study to investigate the effect of food on the relative bioavailability of a 2.5 mg linagliptin+1000 mg metformin fixed dose combination (FDC) tablet

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria: based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
2. Age 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR, and ECG) which deviated from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy), psychiatric disorders, or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells, or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs within 1 month or less than 10 half-lives of the respective drug prior to first study drug administration
10. Participated in another trial with an investigational drug within 2 months prior to administration or during the trial
11. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes daily)
12. Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
13. Drug abuse
14. Blood donation (more than 100 mL within 4 weeks prior to administration)
15. Any laboratory value outside the reference range that was of clinical relevance
16. Inability to comply with dietary regimen of trial site

    For female subjects of childbearing potential only:
17. Positive pregnancy test, pregnancy, or had planned to become pregnant during the study or within 2 months after study completion
18. No adequate contraception during the study and until 1 month after study completion, e.g. not any of the following: implants, injectables, combined hormonal contraceptives, hormonal intrauterine device, sexual abstinence for at least 1 month prior to first study drug administration, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilization (including hysterectomy). Women who did not have a vasectomised partner, were not sexually abstinent, or were not surgically sterile were asked to use an additional barrier method (e.g. condom)
19. Lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
AUC0-72 (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 to 72 h) | up to 72 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of metformin in plasma over the time interval from 0 h extrapolated to infinity) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 h extrapolated to infinity) | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
AUCt1-t2 (area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | up to 72 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
λz (terminal elimination rate constant in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Number of subjects with clinically significant findings in vital signs | up to 7 days after drug administration
  blood pressure, pulse rate
Number of subjects with clinically significant findings in ECG | up to 7 days after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 7 days after drug administration
Number of subjects with adverse events | up to 7 days after drug administration
Assessment of tolerability by the investigator on a 4-point scale | up to 7 days after drug administration